CLINICAL TRIAL: NCT02945111
Title: Watching Live VIA/VILI Examinations on a Digital Screen May Reduce Patients' Anxiety: a Randomized Trial of an Educational Intervention
Brief Title: Watching Live VIA/VILI Examinations on a Digital Screen May Reduce Patients' Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Patrick Petignat (Other)
Responsible Party: Sponsor-Investigator, Prof. Patrick Petignat, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PB_2016-01745
Record Dates: First submitted 2016-10-18; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Cancer; Anxiety
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-time view (Experimental): Women undergoing Visual Inspection with Acetic Acid (VIA) and Lugol's Iodine (VILI) will watch the cervical images taken throughout the examination in real-time on a digital screen. The patients' anxiety level both before and after the examination will be measured using the Spielberg's State Anxiety Inventory.
  Interventions: Behavioral: Real-time view
- No visual support (Active Comparator): Women in this arm will undergo Visual Inspection with Acetic Acid (VIA) and Lugol's Iodine (VILI) without any visual support. Their anxiety level both before and after the examination will be measured using the Spielberg's State Anxiety Inventory.
  Interventions: Behavioral: No visual support

INTERVENTIONS:
Behavioral: Real-time view
  Arms: Real-time view
Behavioral: No visual support
  Arms: No visual support

SUMMARY:
The purpose of this study is to assess whether the degree of anxiety experienced by women undergoing visual inspection with acetic acid (VIA) and Lugol's iodine (VILI) can be reduced by watching the procedure in real-time on a digital screen.

DETAILED DESCRIPTION:
The study took place in the District of Dschang, Cameroon. Women aged between 30 and 49 years, addressed to undergo a pelvic examination with VIA and VILI, were invited to participate. Throughout the examination, one part of the women underwent the routine VIA/VILI, with no visual support (control group), whereas the other part of patients were shown the pictures of the cervix in real-time on a digital screen (study group). At the end of the procedure, all women had the possibility to see the pictures retrospectively. Randomization determined the women's distribution between the two groups. Their anxiety level was measured by asking them to complete the Spielberg's State Anxiety Inventory (STAI) both prior to and immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in a cervical cancer screening campaign organized by the District hospital of Dschang
* Women understanding the study procedure and accepting voluntarily to participate by signing an informed consent form (ICF).

Exclusion Criteria:

* Women not able to comply with the study protocol.

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Within thirty minutes of the VIA/VILI examination
  Anxiety level will be assessed through the STAI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Dschang District Hospital, Dschang, Yaoundé, Cameroon

REFERENCES:
- [Derived] Camail R, Kenfack B, Tran PL, Viviano M, Tebeu PM, Temogne L, Akaaboune M, Tincho E, Mbobda J, Catarino R, Vassilakos P, Petignat P. Benefit of Watching a Live Visual Inspection of the Cervix With Acetic Acid and Lugol Iodine on Women's Anxiety: Randomized Controlled Trial of an Educational Intervention Conducted in a Low-Resource Setting. JMIR Cancer. 2019 May 13;5(1):e9798. doi: 10.2196/cancer.9798. PMID 31094335